CLINICAL TRIAL: NCT05449392
Title: Topical Antibacterial Agents for Prevention of COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2000032248; INV-038276 (Other Grant/Funding Number: Gates Foundation)
Record Dates: First submitted 2022-07-06; First posted 2022-07-08 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: COVID-19; SARS-CoV2 Infection
Keywords: Neosporin; Antibacterial agent; intranasal application
MeSH Terms: conditions — COVID-19 | interventions — bacitracin zinc, neomycin sulfate, polymyxin B, drug combination; Petrolatum

STUDY DESIGN:
Intervention Model Description: Run-in cohort to test optimal sampling and storage conditions: For 6 participants, the investigator will test 50:50 with Neosporin vs Placebo participant nasal sampling and shipping protocol to evaluate signal to noise of interferon-stimulated genes (ISG) measures. If needed, we will rerun the power calculations.
Who Masked: Participant, Investigator
Masking Description: Blinding will be achieved by masking and packaging the products in an identical fashion. Investigational product will be filled in empty Aluminum Ointment Tubes 15 g (Supplied via HealthCareLogistics, Item # 10201-01). The empty Aluminum Ointment Tubes are sterilized by gamma irradiation and have protective inner (epoxy phenolic) coating to prevent ointments from sticking to the sides and reacting with the aluminum.
  Each tube will be filled with approximately 15 g of the Neosporin ointment investigational product, or Vaseline Petroleum Jelly its matching placebo, and labeled in a blinded fashion.
  Patient or clinicians requesting unblinding will contact the principal investigator (PI).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neosporin (Experimental): Neosporin will be distributed by the Yale Investigational Pharmacy. Subjects are to use Neosporin twice a day for 7 days.
  Interventions: Drug: Neosporin
- Vaseline or equivalent (Placebo Comparator): Vaseline or equivalent will be distributed by the Yale Investigational Pharmacy. Subjects are to use Vaseline twice a day for 7 days.
  Interventions: Other: Vaseline

INTERVENTIONS:
Drug: Neosporin — Neosporin is neomycin, bacitracin and polymyxin B with formulation 3.5mg/400 units/5,000 units. The subject will self-apply a small amount (approximately 0.5 g) of the ointment topically into each nostril (intranasal) twice daily (morning and evening) for seven days. Subjects are to pinch the nose to spread the cream.
  Arms: Neosporin
Other: Vaseline — The subject will self-apply a small amount (approximately 0.5 g) of the ointment topically into each nostril (intranasal) twice daily (morning and evening) for seven days. Subjects are to pinch the nose to spread the cream.
  Arms: Vaseline or equivalent

SUMMARY:
The primary objective of this study is to determine whether intranasal application of aminoglycoside (Neosporin) increases local nasal innate immune responses compared to placebo control in healthy participants.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether intranasal application of aminoglycoside (Neosporin) increases local nasal innate immune responses compared to placebo control in healthy participants.

This study will evaluate the role of nasally applied neomycin at inducing local antiviral interferon responses that have been associated with protection against SARS-CoV2 ( severe acute respiratory syndrome coronavirus 2). Local interferon immune responses including the nasal compartment are important in driving early protective responses against the virus. Given the current challenges with vaccine access in lower- and middle-income countries (LMIC) as well as varying vaccine acceptance and hesitancy, additional strategies are needed to help curb the spread of SARS-CoV2. There is a need for easily available agents that are low cost and effective at decreasing the effects of SARS-CoV2 exposure. The investigators will evaluate the effectiveness of intranasal Neosporin (which contains neomycin) at inducing interferon responses in human subjects.

This will be a proof of concept that such approach will provide local immune response that could be beneficial against the SARS-CoV2 infection. The potential impact of this study is the utilization of existing and available topical medications for the purpose of providing local prophylaxis against SARS-CoV2.

The overall hypothesis is that neomycin containing agents such as Neosporin when applied topically in the nose can induce local antiviral interferon responses in adult human subjects. Neosporin will be compared to placebo, control Vaseline (Unilever) or equivalent. A run-in cohort of 6 participants to test optimal sampling and storage conditions will be used. The focus of this study is the randomized double-blinded placebo-controlled trial.

The study will enroll an estimated 40 healthy subjects at one study site, Yale University. Local nasal immune responses will be measured using RT-PCR and multiplex ELISA for interferon response. Participants will apply a small amount of the cream (less than a pea size) to the inside of both nostrils, then pinch the nose to spread the cream. Participants will use Neosporin or placebo twice a day for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Completion of written informed consent
* Covid-negative within 48 hours of enrollment based on PCR or Antigen test. If subjects are found to be positive, the PI will recommend appropriate follow-ups.
* In good general health as evidenced by medical history
* Ability to take Nasal medication and be willing to adhere to the nasal agent regimen

Exclusion Criteria:

* Participant with active nasal or respiratory symptoms.
* Participant with active or chronic respiratory nasal or respiratory infections and or is currently on antibiotics
* Participant who has been treated with oral or topical antibiotics with the past 14 days
* Participant who is on intranasal or oral corticosteroids or systemic immunosuppression medication
* Participant who has immunocompromised conditions such as rheumatological diseases, HIV, cancer on chemotherapy or biologic therapies.
* Participant who is on any intranasally applied medications (prescription or over the counter) including nonmedical nasal products and the use of Netipot or other nasal flush products.
* Participant with known allergic history to Neosporin (allergic history to neomycin or bacitracin or polymyxcin or pramoxine or the inactive ingredients that include cocoa butter, cottonseed oil, olive oil, sodium pyruvate, tocopheryl acetate and white petrolatum)
* Participant with known allergies to aminoglycoside antibiotics (neomycin, tobramycin, gentamycin, others)
* Participant with history of COVID-19 infection in the past 8 weeks.
* Participant who is pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Change in in interferon response profile from nasal samples collected measured by a multiplex ELISA assay | From baseline up to Month 1
  Measurement of interferon response from samples collected using a multiplex ELISA to detect which interferon-stimulated genes (ISGs) are present in sample. ISGs measured include Irf7, Oas1a, Oasl2, Cxcl9, and CxcL10 as well as other corresponding interferons such as Ifna, ifnb, and ifnl
Change in in interferon response gene expression profile from nasal samples collected measured by RT-PCR | From baseline up to Month 1
  Measurement of interferon response from samples collected using RT-PCR to detect expression of ISGs. ISGs measured include Irf7, Oas1a, Oasl2, Cxcl9, and CxcL10 as well as other corresponding interferons such as Ifna, ifnb, and ifnl
Change in RNA expression profile of ISGs using RNAseq assay | Day 1and Day 8
  In a subset of subjects in both arms, RNAseq will be performed to assess the presence and quantity of RNA on samples collected at Day 1 and Day 8. ISGs assessed include Irf7, Oas1a, Oasl2, Cxcl9, and CxcL10 as well as other corresponding interferons such as Ifna, ifnb, and ifnl
Change in RNA expression profile of ISGs using single cell RNAseq assay | Day 1 and Day 8
  In a subset of subjects in both arms, single cell RNAseq will be performed to assess the presence and quantity of RNA on single cells from samples collected at Day 1 and Day 8. ISGs assessed include Irf7, Oas1a, Oasl2, Cxcl9, and CxcL10 as well as other corresponding interferons such as Ifna, ifnb, and ifnl

CONTACTS AND LOCATIONS:
Overall Officials: Charles Dela Cruz, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes